CLINICAL TRIAL: NCT02620397
Title: Clinical Study to Validate the Use of a New Point of Care Troponin I Test as an Aid in the Diagnosis of Myocardial Infarction and Prognosis of Subjects Presenting With Symptoms of Acute Coronary Syndrome
Brief Title: Clinical Study to Validate the Use of a New Point of Care Troponin I Test
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Trinity Biotech (Industry)
Responsible Party: Sponsor
Other Study IDs: CP7001_5ACS
Record Dates: First submitted 2015-11-27; First posted 2015-12-03 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA Whole Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This trial is designed as a prospective, multi-center, observational study of "all-comers" eligible adult subjects presenting to participating emergency departments with symptoms suggestive of acute coronary syndrome (ACS)

DETAILED DESCRIPTION:
This trial is designed as a prospective, multi-center, observational study of "all-comers" eligible adult subjects presenting to participating Emergency Departments (EDs) with symptoms suggestive of ACS and/or myocardial ischemia. Subjects presenting with symptoms suggestive of ACS will be screened and approached for consent for study enrollment by trained personnel.

After obtaining written informed consent, subjects will have up to 4 blood samples collected for cTnI testing using the Meritas Troponin I test and Meritas point-of-care (POC) Analyzer. Blood draws and testing will occur at 4 intervals over 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent must be signed by the subject, or the subject's legal authorized representative.
2. 21 years of age or greater at the time of enrollment
3. Subjects presenting to the ED with any symptoms suggestive of ACS and/or myocardial ischemia, such as but not limited to: subjects currently having chest pain, pressure or a burning sensation across the precordium and epigastrium, pain that radiates to neck, shoulder, jaw, back, upper abdomen and either arm.

Exclusion Criteria:

1. Informed consent form not signed
2. Age <21 years
3. Known pregnancy -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 1000 to 1500 adult subjects presenting to emergency departments (ED) with symptoms suggestive of acute coronary sydrome (ACS) and/or myocardial ischemia
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of the Meritas Troponin I test | 24-hours
  Clinical performance indicators (Sensitivity, Specificity, Positive Predictive Value (PPV) and Negative Predictive Value (NPV) and their respective 95 % confidence intervals (CIs) will be calculated for the quantitative determination of cardiac troponin I (cTnI) for use as an aid in the diagnosis of myocardial infarction (MI)

SECONDARY OUTCOMES:
Prognostic capability of sponsor's Meritas Troponin I to predict mortality (all-cause death) and cardiac events (i.e., MI, cardiac death). | 1 year
  Kaplan-Meier survival curves and risk ratios. A multivariate Cox proportional model with known risk factors as covariates in addition to the Troponin test result will be included in the data analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jim Rock, Study Director — Trinity Biotech
Locations (14):
- United States (14):
  - San Francisco General Hospital & Trauma Center, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Eastern Idaho Regional Medical Center, Idaho Falls, Idaho
  - Kentucky Clinical Trials Laboratories, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Hennepin County Medical Ctr, Minneapolis, Minnesota
  - Sunrise Hospital, Las Vegas, Nevada
  - Carolinas Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Thomas Jefferson Univeristy, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Ben Taub, Houston, Texas